CLINICAL TRIAL: NCT03487731
Title: A Phase I/II, Randomized, Blinded and Placebo-controlled Trial to EValuate the Safety and Potential Efficacy of Allogeneic Human Mesenchymal Stem Cell Injection in PAtieNts With FaceTogenic Back Pain
Brief Title: Allogeneic Human Mesenchymal Stem Cell Injection in PAtieNts With FaceTogenic Back Pain
Acronym: VALIANT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI decided to not proceed with study
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Study Sponsor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180018
Record Dates: First submitted 2018-03-13; First posted 2018-04-04 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Facetogenic Back Pain; Back Pain
Keywords: stem cells; back pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Placebo (Placebo Comparator): Group 1 - Five (5) subjects will be treated with a single administration of 1 cc of 1% lidocaine with 1 cc of 2% Ropivicaine and 0.5 cc of betamethasone soluspan (celestone) solution delivered via intra-facet injection. These subjects will be part of the control (Standard care) group.
  Interventions: Drug: Placebo
- Group 2 - Allogeneic Human Mesenchymal Stem Cells (hMSCs) (Experimental): Group 2 - Five (5) subjects will be treated with a single administration of 20 million allogeneic mesenchymal stem cell delivered intra-facet via 6 injections of 1.5 mL per injection, total of 9 to 12ml. These subjects will be part of the experimental group.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (hMSCs)
- Group A - Allogeneic Human Mesenchymal Stem Cells (hMSCs) (Experimental): Group A will consist of 15 subjects that will receive 20 million Allogeneic hMSCs delivered via lumbar level injection based on pain originator.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (hMSCs)
- Group B - Placebo (Placebo Comparator): Group B will consist of 15 subjects who will receive 2% Ropivicaine and 0.5 cc of betamethasone soluspan (celestone) solution via lumbar level injection based on pain originator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Allogeneic Human Mesenchymal Stem Cells (hMSCs) — A single administration of 20 million allogeneic mesenchymal stem cell delivered intra-facet via 6 injections of 1.5 mL per injection, total of 9 to 12ml.
  Other Names: allo-hMSCs; stem cells
  Arms: Group 2 - Allogeneic Human Mesenchymal Stem Cells (hMSCs); Group A - Allogeneic Human Mesenchymal Stem Cells (hMSCs)
Drug: Placebo — A single administration of 1 cc of 1% lidocaine with 1 cc of 2% Ropivicaine and 0.5 cc of betamethasone soluspan (celestone) solution delivered via intra-facet injection.
  Arms: Group 1 - Placebo; Group B - Placebo

SUMMARY:
The study is a phase I/II trial where allogeneic human mesenchymal stem cells (hMSCs) are injected intracfect into the lumbar facet joints. Forty (40) subjects are scheduled to undergo injection after meeting all inclusion/exclusion criteria will be evaluate at baseline.

DETAILED DESCRIPTION:
There are 40 subjects that will be randomized into the trial into one of 4 groups. In the pilot phase 5 subjects will be enrolled into Group 1, and another 5 subjects will be enrolled into Group 2. Subjects in group 1 will receive placebo but will be eligible for a cross over phase where they will receive a injection of the study investigational product.

In the pilot phase, the first three (3) subjects in each treatment group will not be treated less than 10 days apart.

Following the pilot study, thirty (30) subjects will be scheduled to undergo CT guided facet injection of the lumbar facet joints using a posterior approach after meeting all inclusion/exclusion criteria and baseline evaluation.

Eligible participants will be randomized to either Group A or Group B.Group A will consist of 15 subjects that will receive 20 million Allogeneic hMSCs. Group B will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must:

1. Provide written informed consent.
2. Subjects age >18 and <75 years at the time of signing the Informed Consent Form.
3. Facetogenic back pain diagnosed using the following diagnostic criteria:

   * The facet joint may be affected by systemic disease, as rheumatoid arthritis and ankylosing spondylitis, or be site of micro traumatic fractures, osteoarthritis, meniscoid entrapment, synovial impingement, joint subluxation, synovial inflammation, loss of cartilage, and mechanical injury.
   * Pain onset at dorsal extension and release at flexion is often considered suggestive for facet pain, even if non-specific, such as maximal tenderness upon deep palpation of posterior elements
   * History of temporary improvement with a medial branch block anesthetic injection of the targeted joints
   * Axial lumbar pain without radicular symptoms
   * Pain on hyperextension, rotation, and lateral bending with physical exam
4. Chronic facetogenic pain (≥ 6 months) in patients that have failed conservative management. (This includes but is not limited to a trial of oral medications, 6 weeks of physical therapy, intra-articular injection of the facet joints, and/or facet joint medial branch neurotomy.)
5. Diagnosis of lumbar facet joint pain confirmed by analgesic injections.
6. Have spinal level L3-4, L4-5 and L5-S1 bilaterally for bilateral pain and same side only for unilateral pain.

Exclusion Criteria:

In order to participate in this study, a subject must not:

1. Previous surgical intervention for back pain
2. Previous mesenchymal stem cell (MSC) injection(s) in to facet joints
3. Use of anticoagulation or NSAIDs within 5 days of the injection
4. MRI finding of severe high grade lumbar stenosis
5. Leg pain exceeding back pain
6. Pain worse with flexion maneuvers
7. Fracture of lumbar vertebrae
8. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.
9. Inability to perform any of the assessments required for endpoint analysis.
10. Clinically abnormal screening laboratory values.
11. Serious comorbid illness or any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
12. Hypersensitivity to dimethyl sulfoxide (DMSO).
13. Be an organ transplant recipient.
14. Have a clinical history of malignancy within 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma, if recurrence occurs.
15. Have a non-pulmonary condition that limits lifespan to < 1 year.
16. Have a history of drug or alcohol abuse within the past 24 months.
17. Be serum positive for HIV, hepatitis BsAg or Viremic hepatitis C.
18. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of any treatment-emergent serious adverse events | at one-month post injection
  Incidence (at one-month post injection) of any treatment-emergent serious adverse events.

SECONDARY OUTCOMES:
Difference in subject quality of life assessment - SF-12 | Baseline, Month 3, and Month 6
  Difference in subject quality of life assessment - SF-12 to assess if there is improvement in health via this health survey.
Difference in subject quality of life assessment - Oswestry Low Back Pain | Baseline, Month 3, and Month 6
  Difference in subject quality of life assessment - Oswestry Low Back Pain where the scores are defined by percentage with 0 to 20% showing minimal disability and 81-100% showing severe disabling symptoms.
Death from any cause. | Baseline, Month 3, and Month 6
  Death from any cause.
Change in pain using the Numeric rating scale | Baseline and Month 6
  Change between baseline and 6 months in pain using the Numeric Rating Scale (NRS) scale. This is assessed on a scale from 0 to 10 with 0 being no pain and 10 being the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sherman, MD, Principal Investigator — University of Miami
Locations (1):
- ISCI / University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute website — http://ISCI.med.miami.edu